CLINICAL TRIAL: NCT06569420
Title: A Randomized, Multicenter, Phase III Open-label Study: Efficacy and Safety of Comparing SAF-189s With Crizotinib in First-line Anaplastic Lymphoma Kinase-positive Advanced and Metastatic NSCLC
Brief Title: Study Of Comparing SAF-189s With Crizotinib In First Line ALK-Positive Advanced and Metastatic NSCLC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAF-189-III101
Record Dates: First submitted 2024-08-02; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Non-Small Cell Lung Cancer; ALK-positive; SAF-189s
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foritinib Succinate (Experimental): Foritinib Succinate capsules will be administered orally at a dose of 160 mg QD until disease progression, unacceptable toxicity withdrawal of consent, or death.
  Other Names: SAF-189s
  Interventions: Other: Drug: Foritinib Succinate
- Control: Crizotinib (Active Comparator): Crizotinib capsules will be administered orally at a dose of 250 mg BID until disease progression, unacceptable toxicity withdrawal of consent, or death.
  Interventions: Other: Drug: Crizotinib

INTERVENTIONS:
Other: Drug: Foritinib Succinate — SAF-189s: 160 mg QD, 21 days a cycle
  Other Names: SAF-189s
  Arms: Foritinib Succinate
Other: Drug: Crizotinib — Crizotinib: 250 mg BID, 21 days a cycle
  Arms: Control: Crizotinib

SUMMARY:
This randomized, multicenter, Phase III, open-label study will evaluate the efficacy and safety of SAF-189s versus crizotinib treatment in participants with treatment-naive ALK-positive advanced NSCLC. Participants will be randomized 1:1 into one of the two treatment groups to receive either SAF-189s (160 milligrams [mg] once daily [QD]) or crizotinib (250 mg BID) orally, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Sufficiently understand the study and are willing to sign the informed consent form (ICF);
* Male or female patients ≥ 18；
* Histologically or cytologically confirmed diagnosis of local advanced (Stage IIIB/IIIC) or metastatic (Stage IV) NSCLC;
* ALK-positive as assessed by the Ventana immunohistochemistry (IHC) test. Sufficient tumor tissue available to perform ALK IHC is required. Ventana IHC testing will be performed at the designated central laboratory;
* Measurable disease by response evaluation criteria in solid tumors (RECIST) version 1.1 (v1.1) prior to the administration of study treatment; Lesions that have received radiation therapy cannot be considered as target lesions unless there is confirmed progression of the lesion after radiation therapy;
* Participants with no prior systemic treatment for local advanced (Stage IIIB/IIIC not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC;
* Eastern cooperative oncology group performance status (ECOG PS) of 0-2;
* Life expectancy of at least 12 weeks;
* Adequate organ and bone marrow function as documented by:Hematologic function: absolute neutrophil count (ANC) ≥1.5 × 10^9/L; hemoglobin≥ 90 g/L; Platelet count ≥ 100 × 109/L;Serum total bilirubin ≤ 1.5 × ULN (if the patient has Gilbert's syndrome, ≤ 3 × ULN and direct bilirubin ≤ 1.5 × ULN);Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for patient with liver metastases);Creatinine clearance (CrCL) ≥ 50 mL/min (calculated by Cockcroft-Gault equation)；Baseline QTc ≤470 ms corrected by Fridericia fomula;Baseline LVEF≥50%;
* For all females of childbearing potential (FCBP), a negative serum pregnancy test result must be obtained within 7 days prior to starting study treatment, and agree to use a highly effective method of contraception, during the treatment period and for 3 months following the last dose of study drug.For men whose partners are fertile women, agreement to remain abstinent or use a condom plus an additional contraceptive method during the treatment period and for at least 3 months after the last dose of study drug. Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. This protocol defines a FCBP as a sexually mature woman who:1）has not undergone a hysterectomy or bilateral oophorectomy；2）has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out child-bearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Has had prior anti-cancer treatment with biological drugs, or other investigational agents within 28 days; or received chemotherapy, TKI or targeted therapies within 14 days prior to enrollment; or based on the last administration within 5 half-life of the drug (whichever is shorter);
* Patients with central nervous system (CNS) metastases requiring: 1）clinical local intervention such as surgical excision, radiotherapy or other therapies (known brain metastasis or other CNS metastasis that is either asymptomatic or symptomatic but requiring no local interventions may qualify for the study per the investigator); 2）patients requiring systemic treatment with corticosteroids and >10 mg/day prednisone or equivalent; 3）requiring antiepileptic drug sustained treatment;
* Spinal cord meatstasis with potential risk of or symptomic spinal cord compression;
* National cancer institute common terminology criteria for adverse events (NCI CTCAE) (version 5.0) Grade 2 or higher toxicities due to any prior therapy (e.g., chemotherapy, surgery or radiotherapy) (excluding alopecia)
* Patient has uncontrolled diabetes and intervented by insulin (patient with fasting blood glucose levels <9.8 mmol/L under stable oral hypoglycemic medications allowed to be enrolled);
* Has a history of acute pancreatitis within 1 year before enrollment, ;
* Patients have history of interstitial lung disease, drug-induced interstitial lung disease or induced by radiation therapy and requring hormone therapy, or still receiving medication or other clinical intervention, or currently having active pulmonary interstitial lesions;
* The patients had uncontrollable amounts of pleural effusion, ascites, and pericardial effusion.
* Patients with inability to swallow or with active digestive system disease or underwent major GI surgery, which remarkably affect oral administration or absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea and vomiting, diarrhea, malabsorption syndrome, and small bowel resection);
* History of hypersensitivity to any of the additives in the SAF-189s and drug formulation;
* History of hypersensitivity to any of the additives in the crizotinib and drug formulation;
* Patients with clinically significant active bacterial, fungal or viral infections, including hepatitis B virus surface antigen-positive and hepatitis B virus DNA over 2000 IU/mL, positive for hepatitis C virus (HCV) antibody test; confirmed human immunodeficiency virus (HIV) infection, and those who are unwilling to undergo HIV testing; hepatitis B carriers are allowed to be enrolled;
* Patients have other malignant tumor history in 3 years or with other malignant tumors simultaneously (excluding curatively treated in situ carcinoma of cervix cancer, non-melanoma skin basal cell carcinoma, thyroid carcinoma in situ, and any cured tumor which is considered to have no impact in progression-free survival (PFS) or overall survival (OS) for the current NSCLC);
* Patients with cardiac function impairment or clinically significant heart diseases, including congestive heart-failure New York Heart Association (NYHA) III or above, arrhythmias (including but not limited to complete left bundle branch Atrioventricular block complete and atrioventricular block second degree), conduction abnormality requiring medication, severe coronary artery disease, heart valve disease or myocardiopathy or uncontrolled hypertension;
* Patients who received major surgery within 3 weeks before enrollment or have not adequately recovered from prior surgery. Major surgery is defined as Grade 3 or 4 surgery per Management Measures for Clinical Application of Medical Technology implemented on May 1st, 2009 in China;
* Patients who have been received one of the following treatments: 1）strongly inhibits or induces of CYP3A4, repaglinide (cytochrome [CYP]2C8 sensitive substrate) and drugs metabolized via CYP3A4 enzyme within 1 week before enrollment; 2）medicines which are known to cause QT prolongation or torsade de pointes;3）coumarin anticoagulants within 1 week before enrollment (low molecular weight heparin is permitted);4）illegal drugs;
* Pregnant or lactating: any subjects who experience pregnancy during the trial need to withdraw from the study.
* Any other clinically significant disease or condition, or acute or chronic medical conditions (such as uncontrolled diabetes), or mental condition or abnormal lab test, that investigator assesses that maybe increase the risk of participating or affect the interpretation of research reslults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by IRC | up to 36 months
  as determined by IRC based on RECIST 1.1 criteria.
Overall survival (OS) | up to 60 months
  Time in months from date of randomization to death due to any cause
Progression-free survival (PFS) by INV | up to 36 months
  as determined by INV based on RECIST 1.1 criteria.
Objective Response Rate (ORR) by IRC and INV | up to 36 months
  Percentage of Participants With Objective Response Rate (ORR) of Complete Response (CR) or Partial Response (PR) as Determined by Investigators and IRC According to RECIST V1.1 Criteria
Duration of response (DOR) by IRC and INV | up to 36 months
  Duration of response defined as time from when response was first documented until first documented disease progression or death, whichever occurs first.
to evaluate the C-ORR in patient with CNS metastases. | up to 36 months
to assess the C-TTR in patient who have as CNS objective response | up to 36 months
to assess the C-DOR in patient who have as CNS objective response. | up to 36 months
to assess the C-TTP in patient who have as CNS objective response. | up to 36 months
The time to CNS progression in ITT by IRC. | up to 36 months
  To evaluate the time to CNS progression in ITT by IRC.
Incidence of adverse events. | up to 36 months
Health-Related Quality of Life (HRQoL) by EORTC Quality of Life Questionnaire C30 Score | up to 36 months
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a better level in functional scales/items and Global health status, or worse level in symptom scales/items.
Health-Related Quality of Life (HRQoL) by EORTC Quality of Life Questionnaire LC13 Score | up to 36 months
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a worse level in symptom scales/items, such as in cough, short breath, chest pain, and other symptoms associated with lung cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No